CLINICAL TRIAL: NCT01133275
Title: A Phase II Clinical Trial of Lenalidomide and Prednisone in Low and Intermediate-1 IPSS Risk, Non-del (5q) MDS Patients
Brief Title: Lenalidomide and Prednisone in Low and Int-1 Myelodysplastic Syndrome (MDS) Non 5q MDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16099; RV-MDS-PI-0456 (Other: Celgene Corp.); 25005/1 (Other: Quorum Review IRB)
Record Dates: First submitted 2010-05-25; First posted 2010-05-28 (Estimated); Results first posted 2016-01-18 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Myelodysplastic Syndrome; MDS
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Prednisone; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lenalidomide and Prednisone Therapy (Experimental): All participants received lenalidomide and prednisone therapy for 6 cycles (24 weeks). Each cycle is 28 days (4 weeks).
  Interventions: Drug: Prednisone; Drug: Lenalidomide

INTERVENTIONS:
Drug: Prednisone — Prednisone therapy for 6 cycles (24 weeks).
  Other Names: Deltasone
Drug: Lenalidomide — Lenalidomide therapy for 6 cycles (24 weeks).
  Other Names: REVLIMID®

SUMMARY:
The purpose of this research is to evaluate the use of lenalidomide and prednisone in people with Myelodysplastic Syndrome (MDS).

Lenalidomide is a drug that alters the immune system and it may also interfere with the development of tiny blood vessels that help support tumor growth. Therefore, in theory, it may reduce or prevent the growth of cancer cells. Lenalidomide is approved by the U.S. Food and Drug Administration (FDA) for the treatment of specific types of myelodysplastic syndrome (MDS) and in combination with dexamethasone for people with multiple myeloma (MM) who have received at least 1 prior therapy. MDS and MM are cancers of the blood. It is currently being tested in a variety of cancer conditions. As it is being used in this study it is considered an investigational use. An "investigational use" is a use that is being tested and is not approved by the FDA.

Prednisone is approved by the FDA to treat numerous conditions. In addition, prednisone is approved by the FDA to treat Low or Intermediate-1 IPSS Risk, non-del (5q) MDS.

"Study drug" refers to the combination of lenalidomide and prednisone.

DETAILED DESCRIPTION:
10 mg/day of lenalidomide will be taken by mouth on days 1 - 28 of cycles 1-6. Dosing will be in the morning at approximately the same time each day.

Planned prednisone dose:

* 30 mg by mouth daily, days 1-28 of cycle 1
* 20 mg by mouth daily, days 1-28 of cycle 2
* 10 mg by mouth daily, days 1-28 of cycle 3
* 10 mg by mouth every other day on days 1-28 of cycles 4-6
* 5 mg by mouth every other day for responders beyond cycle 6

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form
* Age ≥ 18 years at the time of signing the informed consent form
* Able to adhere to the study visit schedule and other protocol requirements
* Documented diagnosis of MDS according Word Health Organization (WHO) that meets International Prognostic Scoring System (IPSS) criteria for Low- to Intermediate-1-risk disease or non-proliferative (white blood count [WBC] < 13,000/uL) chronic myelomonocytic leukemia (CMML) and MDS/myeloproliferative neoplasms (MPN).
* Absence of a chromosome 5q deletion by metaphase cytogenetics or fluorescent in situ hybridization (FISH) analysis
* Red blood cell (RBC) transfusion-dependent anemia defined as having received ≥4 transfusions of RBCs for hemoglobin (Hgb) ≤ 9.0 g/dl within 56 days of randomization or symptomatic anemia (Hgb ≤ 9.0 g/dl)
* No response or progression on prior treatment with epoetin alpha (> 40,000 U/wk x 6), darbepoetin alpha (≥ 500 mcg q 3 wk x 2) or serum erythropoietin (EPO) concentration ≥ 500 mU/ml
* All previous cancer therapy, including radiation, hormonal therapy and surgery, must have been discontinued at least 4 weeks prior to treatment in this study.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2 at study entry
* Laboratory test results within these ranges: Absolute neutrophil count ≥ 500 /mm³; Platelet count ≥ 50,000 /mm³; Creatinine Clearance > 60 mL/min by Cockcroft-Gault formula; Total bilirubin ≤ 1.5 mg/dl; aspartic transaminase (AST)and alanine transaminase (ALT) ≤ 2 x upper limit of normal (ULN).
* Disease free of prior malignancies for ≥ 3 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "insitu" of the cervix or breast
* Must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 milli-international units per milliliter (mIU/mL) within 10 - 14 days prior to and again within 24 hours of prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from signing the informed consent form.
* Pregnant or breast feeding. (Lactating females must agree not to breast feed while taking lenalidomide).
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy within 28 days of baseline
* Known hypersensitivity to thalidomide
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs or history of desquamating (blistering) rash while taking thalidomide
* Any prior use of lenalidomide
* Concurrent use of other anti-cancer agents or treatments
* Known positive for human immunodeficiency virus (HIV) or infectious hepatitis, type B or C
* Proliferative CMML (WBC ≥13,000/μL)
* MDS secondary to treatment with radiotherapy, chemotherapy, and/or immunotherapy for malignant or autoimmune diseases
* Prior ≥ grade-2 National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) allergic reaction to thalidomide
* Clinically significant anemia due to factors such as iron, B12 or folate deficiencies, autoimmune or hereditary hemolysis or gastrointestinal bleeding
* Known HIV-1 positivity
* Chromosome 5q deletion
* Documented thromboembolic event within the past 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-04-28 (Actual); Primary Completion 2015-01-31 (Actual); Study Completion 2019-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rami Komrokji, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- United States (2):
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at Moffitt Cancer Center and Shands Cancer Hospital at the University of Florida from 4/28/2010 through 8/13/2013.
Groups:
- Lenalidomide and Prednisone Therapy: Lenalidomide and prednisone therapy for 6 cycles (24 weeks). Each cycle is 28 days (4 weeks).
Period: Overall Study
Arm/Group | Lenalidomide and Prednisone Therapy
Started | 28
Completed | 26
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Cerebrovascular accident (CVA) | 1

BASELINE CHARACTERISTICS:
Population: All participants
Arm/Group | Lenalidomide and Prednisone Therapy
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 20
Age, Continuous [Mean (Full Range); unit: years] | 68.64 [22 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Erythroid Response
Description: The rate of erythroid response to treatment with the lenalidomide/prednisone combination in non-del (5q) low and int-1 risk Myelodysplastic Syndrome (MDS) with symptomatic anemia. Hematological improvement erythroid response (HI-E) according to International Working Group (IWG) 2006 criteria.
Time Frame: Up to 7 months
Population: All evaluable participants
Measure: Number; unit: participants
Arm/Group | Lenalidomide and Prednisone Therapy
Number analyzed (Participants) | 26
participants | 5

2. Secondary Outcome: Number of Participants With Grade 3 or 4 Adverse Events Possibly Related to Treatment
Description: Grade 3 or 4 events Related/Possibly Related/Probably Related to study treatment. Number of participants with events specified in the study protocol: Neutropenia, Thrombocytopenia, Febrile Neutropenia, Infection, Sepsis, Venous Thromboembolic Events. Evaluations according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) V4.0.
Time Frame: Up to 54 months
Population: All participants
Measure: Number; unit: participants
Arm/Group | Lenalidomide and Prednisone Therapy
Number analyzed (Participants) | 28
participants
  Neutropenia | 8
  Thrombocytopenia | 4
  Febrile Neutropenia | 0
  Infection and Sepsis | 0
  Venous Thromboembolic Events | 0

ADVERSE EVENTS:
Time Frame: 4 years, 6 months
Arm/Group | Lenalidomide and Prednisone Therapy
Serious Adverse Events (participants affected / at risk) | 8/28
Other Adverse Events (participants affected / at risk) | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide and Prednisone Therapy (N=28)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Blood clot (Blood and lymphatic system disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
Heart arrhythmia (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Rectal bleeding (Gastrointestinal disorders) | 1 (1)
Severe abdominal cramping (Gastrointestinal disorders) | 1 (1)
Severe nausea (Gastrointestinal disorders) | 1 (1)
Uncontrolled vomiting (Gastrointestinal disorders) | 1 (1)
Small intestinal blockage (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Sudden death NOS (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Pain - sore throat (General disorders) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Stroke / Cerebrovascular Accident (CVA) (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide and Prednisone Therapy (N=28)
Diarrhea (Gastrointestinal disorders) | 13 (18)
Constipation (Gastrointestinal disorders) | 6 (7)
Nausea (Gastrointestinal disorders) | 5 (7)
Vomiting (Gastrointestinal disorders) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 2 (3)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 13 (14)
Edema limbs (General disorders) | 7 (10)
Paul (General disorders) | 7 (9)
Fever (General disorders) | 5 (5)
Chills (General disorders) | 4 (4)
Platelet count decreased (Investigations) | 16 (37)
Neutrophil count decreased (Investigations) | 13 (49)
White blood cell decreased (Investigations) | 13 (40)
Creatinine increased (Investigations) | 2 (2)
Investigations - Other (Investigations) | 2 (4)
Lymphocyte count decreased (Investigations) | 2 (5)
Weight gain (Investigations) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 15 (36)
Leukocytosis (Blood and lymphatic system disorders) | 5 (5)
Movements involuntary (Nervous system disorders) | 6 (6)
Dizziness (Nervous system disorders) | 4 (5)
Headache (Nervous system disorders) | 4 (4)
Memory impairment (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (3)
Sinus pain (Nervous system disorders) | 2 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 4 (5)
Bruising (Injury, poisoning and procedural complications) | 6 (6)
Fall (Injury, poisoning and procedural complications) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 3 (4)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 2 (6)
Sinusitis (Infections and infestations) | 2 (2)
Insomnia (Psychiatric disorders) | 6 (6)
Blurred vision (Eye disorders) | 4 (4)
Eye disorders - Other (Eye disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
The study was terminated at the end of step one, as no signal of higher response of the combination was observed compared to what was reported on the MDS-002 study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes